CLINICAL TRIAL: NCT01102361
Title: Study of Prostate Cancer Detection With in House Developed Robot
Brief Title: Ultrasound Based Transperineal Robotic Biopsy of the the Prostate
Acronym: BxB
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Prof. Chris Cheng, Singapore General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BioXbot
Record Dates: First submitted 2010-04-11; First posted 2010-04-13 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2006-05

CONDITIONS: Previous Negative Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transperineal Biopsy (Experimental): Biopsy of the prostate using transperineal approach
  Interventions: Procedure: Robotic Transperineal Biopsy

INTERVENTIONS:
Procedure: Robotic Transperineal Biopsy — Saturation biopsy for previous negative patients

SUMMARY:
The objective of the study is to examine the effectiveness and accuracy of the BioXbot in prostate biopsy as opposed to transrectal biopsy. This evaluation of the efficacy of both the procedures is based on:

* Uptake rate
* Peripheral zone reachability
* Needling accuracy
* Procedure execution time
* Post operative discomfort or trauma experienced by patient
* Quality and type of tissue sample extracted
* Adverse and unanticipated side-effects on patient after the procedure and recording any unexpected reactions

DETAILED DESCRIPTION:
The prostate gland is a walnut-sized organ found only in men that encircles the urethra (urine passage) below the urinary bladder. It secretes fluid that is an important component of semen. Prostate cancer is a disease of the prostate gland where malignant tumours cells invade normal prostate tissue and spread to other organs. It is second leading cause of cancer death in men and it is mainly found in men above the age of 50 years.

Prostate biopsy is considered to be the most definitive diagnostic tool for prostate cancer. It is a surgical procedure in which a small sample of tissue is removed from the prostate gland and examined by a pathologist. The procedure normally takes about 15 minutes and is usually performed by the urologist in conjunction with transrectal ultrasound (TRUS). No anesthetic is required. With the help of TRUS, a doctor guides a biopsy gun -- a hand-held device with a spring-loaded, slender needle -- through the wall of the rectum into the area of the prostate gland that appears abnormal. Since the rectal wall is thin, it is possible to place the needle more accurately and with less injury to other tissues. When activated, the needle can remove a slender cylinder of tissue, called a core.

Transrectal ultrasound-guided prostate biopsy has become the standard for obtaining tissue for the histological diagnosis of prostate cancer. On the other hand, transperineal approach is not commonly used worldwide and little data is available on transperineal prostate biopsy.

However, there are some problems with existing system and these include:

* Random Biopsy Sites: Biopsy cores represent only about 0.6% of the prostate in terms of volume. Therefore, without having accurate knowledge of cancer sites, it is unlikely that a random biopsy protocol will yield consistently high cancer detection rates.
* Inaccurate Needling: The biopsy needle may not reach the desired position accurately and quickly under manual control.
* Limited 2D Guidance: The TRUS used for biopsy guidance is 2D ultrasound images. As the biopsy sites are distributed in 3D, it is difficult for the surgeon to imagine the overall picture of the biopsy sites and identify the biopsy site accurately and intuitively.
* Risk Factors: The two primary risks of needle biopsy are severe bleeding and infection of the prostate gland or urinary tract.
* Transrectal Shortfalls: As most of the cancer occurs at the apex area of the prostate, transperineal biopsy is considered having higher chance to get cancer tissue, comparing with the conventional transrectal biopsy. Furthermore, transperineal biopsy is considered "cleaner", as its puncture point is on skin, rather than on rectum.

To assist the surgeon in transperineal biopsy, a device name BioXbot has been designed. BioXbot aims to address the shortfalls of the transrectal method of biopsy and limitations of existing robotic biopsy in order to improve the cancer uptake rate. An ideal design should need no more than 2 operators to complete the procedure comfortable within comparable time with the conventional approach. A motorized needle positioning mechanism may also improve the accuracy in the needling and allow the needle reach any point within the prostate in all scenarios.

BioXbot is a computer based motion control system with software driven gantry mechanism to assist in the positioning of the biopsy gun. It drives a 2D ultrasound probe to obtain a series of 2D images of the prostate which will then be modeled into a 3D view. This 3D visualization gives the surgeon a better idea of the prostate and allows him to plan the biopsy sites more intuitively. The mechanical components precisely align it to allow the clinician to accurately reach the position inside the prostate he wanted to and obtain tissue from there. To improve the usability and the positioning accuracy, as well as reducing the operation time, the positioning of the needle is fully motorized.

ELIGIBILITY:
Inclusion Criteria:

* At least one normal previous prostate biopsy and at least 2 weeks since prior prostate biopsy
* Increasing prostate-specific antigen (PSA) level
* The Investigator has completed a medical history and a physical examination to assure that the subjects meet all study enrollment criteria

Exclusion Criteria:

* Patient with operative risk ASA ( American Society of Anaesthesia) = or > 4
* A history of bleeding disorders/coagulopathy or ongoing treatment for this condition
* Patients with psychiatric diseases or insufficient cerebral function

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2006-05; Primary Completion 2011-01 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Cancer Detection | 2 years
  to detect any undetected cancer in Patietns undergoing saturation biopsy

SECONDARY OUTCOMES:
Accuracy and Repeatability | 6 months
  To be accurate in biopsy position (+/- 2mm) and be able to go back to the same position if patient undergoes treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore, Singapore